CLINICAL TRIAL: NCT01959802
Title: Correlation Between Foveal Cone Outer Segment Tips Line Defect and Visual Acuity After Surgery for Macular Pseudohole
Brief Title: Foveal Cone Outer Segment Tips Line Defect in Macular Pseudohole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor of Ophthalmology, Kyorin University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kyorineye014; Kyorineye014 (Other: Kyorin Eye Center)
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Macular Psudohole
Keywords: Macular pseudohole; Cone outer segment tips line
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrectomy (Other): Vitrectomy for macular pseudo hole
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
Evaluation of recovery in foveal cone outer segment tips line defect and visual acuity after surgery for macular pseudohole

ELIGIBILITY:
Inclusion Criteria:

* The patienst with macular pseudo hole

Exclusion Criteria:

* The patients with follow-up less than 6 months

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Optical coherence tomography | one year
  Anatomical recovery detected with optical coherence tomography after surgery

SECONDARY OUTCOMES:
Visual acuity | one year
  Visual recovery after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan